CLINICAL TRIAL: NCT03779724
Title: The Effects of Isokinetic Exercises on Muscle Strength, Joint Position Sense, and Kinesiophobia in Patients With Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: Isokinetic Exercises in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dr. Melek Aykut Selçuk, Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5070
Record Dates: First submitted 2018-12-11; First posted 2018-12-19 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; isokinetic; exercises; joint position sense; kinesiophobia
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Kinesiophobia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled trial aimed to recruit 50 patients with MS from the physical medicine and rehabilitation clinic of Ankara Training and Research Hospital, Health Sciences University, Ankara, Turkey. Fifty patients who met the inclusion criteria were enrolled in the study. Fifty patients were randomized to two groups: isokinetic exercise (Group 1) (n=25) and home exercise (Group 2) (n=25). Randomization was completed using sequentially numbered, opaque envelopes by the investigator. All patients gave informed consent before the assessment. The outcome measures were assessed initially and at eighth week after the treatment. Group 1 performed isokinetic concentric quadriceps and hamstring strengthening exercises under supervision and Group 2 performed lower extremity muscle strengthening and balance exercises at home.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isokinetic exercise (Experimental): The isokinetic dynamometer (Biodex Multijoint Pro 3) was used for isokinetic exercises. The isokinetic exercise program was implemented over eight weeks, twice a week on non-consecutive days under the supervision of a doctor. The number of repetitions undertaken by the patients over the program were as follows: first week 5 at 60°/s and 10 at 180°/s, second week 10 at 60°/s and 15 at 180°/s, third week 15 at 60°/s and 20 at 180°/s, fourth week 20 at 60°/s and 30 at 180°/s, and in the last four weeks 20 at 60°/s and 40 at 180°/s angular velocities. Each block of 10 repetitions were performed as a set.
  Interventions: Other: exercises
- home exercise (Active Comparator): The patients undertook lower extremity strengthening and balance exercises three times a week for eight weeks without supervision. They started with three repetitions, which was gradually increased to 10-15. The patients were called two times a week to inquire about exercise continuity and encouraged to undertake the recommended exercises.
  Interventions: Other: exercises

INTERVENTIONS:
Other: exercises

SUMMARY:
The investigators evaluated the effects of isokinetic muscle strengthening exercises of the quadriceps and hamstring on muscle strength, joint position sense, pain, kinesiophobia and quality of life in patients with multiple sclerosis.

DETAILED DESCRIPTION:
Objective: To evaluate the effects of isokinetic exercises on muscle strength, knee joint position sense, pain, kinesiophobia, and quality of life in patients with multiple sclerosis.

Design: Randomized controlled trial. Setting: Outpatient clinic. Participants: Fifty patients with multiple sclerosis. Interventions: Fifty patients who met the inclusion criteria were randomized to an isokinetic exercise (n:25) or home exercise programme (n:25). Sequentially numbered opaque envelopes were used for randomization.

Outcome measures: The outcome measures were the peak torque/body mass index of quadriceps and hamstring muscles at 60°/s and 180°/s velocities, the hamstring/quadriceps ratios at the same velocities, absolute angular errors of the 15°, 45°, and 60° and the mean absolute angular error of joint position sense of the less and more affected knees, and the scores of Multiple Sclerosis Quality of Life-54, Visual Analogue Scale, and Tampa Scale of Kinesiophobia.

ELIGIBILITY:
Inclusion Criteria:

* definite relapsing remitting MS and secondary progressive MS diagnosis
* mild and moderate MS determined by Kurtzke Expanded Disability Status Scale (EDSS) scores below 6.5
* a disease duration of more than one year.

Exclusion Criteria:

* having an acute exacerbation within the last three months
* intravenous pulse steroid therapy in the last four weeks
* grade 3-4 spasticity according to the Modified Ashworth Scale
* severe vision impairment
* severe fatigue and depression
* past knee surgery
* other neurologic diseases
* systemic diseases
* pregnancy
* having received an exercise program within the last four weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melek A Selçuk, MD, Principal Investigator — Aksaray University Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Aksaray University Training and Research Hospital, Aksaray
  - Ankara Training and Researc Hospital, Health Sciences University, Ankara

REFERENCES:
- [Background] Yahia A, Ghroubi S, Mhiri C, Elleuch MH. Relationship between muscular strength, gait and postural parameters in multiple sclerosis. Ann Phys Rehabil Med. 2011 May;54(3):144-55. doi: 10.1016/j.rehab.2011.02.004. Epub 2011 Mar 9. English, French. PMID 21493176
- [Background] Robineau S, Nicolas B, Gallien P, Petrilli S, Durufle A, Edan G, Rochcongar P. [Eccentric isokinetic strengthening in hamstrings of patients with multiple sclerosis]. Ann Readapt Med Phys. 2005 Feb;48(1):29-33. doi: 10.1016/j.annrmp.2004.04.005. French. PMID 15664681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This prospective randomized controlled trial aimed to recruit 50 patients with multiple sclerosis from the physical medicine and rehabilitation clinic of Ankara Training and Research Hospital, Health Sciences University, Ankara, Turkey.
Groups:
- Isokinetic Exercise: The isokinetic dynamometer (Biodex Multijoint Pro 3) was used for isokinetic exercises. The isokinetic exercise program was implemented over eight weeks, twice a week on non-consecutive days under the supervision of a doctor. The number of repetitions undertaken by the patients over the program were as follows: first week 5 at 60°/s and 10 at 180°/s, second week 10 at 60°/s and 15 at 180°/s, third week 15 at 60°/s and 20 at 180°/s, fourth week 20 at 60°/s and 30 at 180°/s, and in the last four weeks 20 at 60°/s and 40 at 180°/s angular velocities. Each block of 10 repetitions were performed as a set.
  exercises
- Home Exercise: The patients undertook lower extremity strengthening and balance exercises three times a week for eight weeks without supervision. They started with three repetitions, which was gradually increased to 10-15. The patients were called two times a week to inquire about exercise continuity and encouraged to undertake the recommended exercises.
  exercises
Period: Overall Study
Arm/Group | Isokinetic Exercise | Home Exercise
Started | 25 | 25
Completed | 19 | 21
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isokinetic Exercise | Home Exercise | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.21 (8.81) | 39.95 (12.25) | 39.60 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 6 | 7 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 19 | 21 | 40

OUTCOME MEASURES:

1. Primary Outcome: Isokinetic Muscle Strength Test of the More and Less Affected Knees
Description: The peak torque/body mass index of the quadriceps and hamstring muscles at 60°/s and 180°/s velocities were measured by an isokinetic dynamometer (Biodex Multijoint Pro 3) in Newton/meter. A definite muscle strength value has not been defined. Literally, healthy controls and patients are compared. Higher scores indicate better muscle strength.
Time Frame: At baseline (10 minutes before the start of the treatment) and 8 weeks after start of the treatment
Measure: Mean (Standard Deviation); unit: Newton/meter
Groups:
- Isokinetic Exercise Baseline: The isokinetic dynamometer (Biodex Multijoint Pro 3) was used for isokinetic exercises. The isokinetic exercise program was implemented over eight weeks, twice a week on non-consecutive days under the supervision of a doctor. The number of repetitions undertaken by the patients over the program were as follows: first week 5 at 60°/s and 10 at 180°/s, second week 10 at 60°/s and 15 at 180°/s, third week 15 at 60°/s and 20 at 180°/s, fourth week 20 at 60°/s and 30 at 180°/s, and in the last four weeks 20 at 60°/s and 40 at 180°/s angular velocities. Each block of 10 repetitions were performed as a set.
  exercises
- Isokinetic Exercise After Treatment: the outcome measurements of isokinetic exercises group after the treatment
- Home Exercise Baseline: The patients undertook lower extremity strengthening and balance exercises three times a week for eight weeks without supervision. They started with three repetitions, which was gradually increased to 10-15. The patients were called two times a week to inquire about exercise continuity and encouraged to undertake the recommended exercises.
  exercises
- Home Exercise After Treatment: the outcome measurements of home exercises group after the treatment
Arm/Group | Isokinetic Exercise Baseline | Isokinetic Exercise After Treatment | Home Exercise Baseline | Home Exercise After Treatment
Number analyzed (Participants) | 19 | 19 | 21 | 21
Newton/meter
  60°/s Quadriceps PT/BMI(less affected knee) | 110.48 (37.20) | 141.05 (31.59) | 123.02 (53.80) | 127.83 (54.35)
  60°/s Hamstring PT/BMI(less affected knee) | 69.25 (24.28) | 85.87 (21.00) | 72.85 (29.02) | 78.40 (31.21)
  60°/s hamstring/quadriceps(less affected knee) | 0.63 (0.14) | 0.61 (0.12) | 0.61 (0.14) | 0.62 (0.12)
  180°/s Quadriceps PT/BMI(less affected knee) | 59.87 (24.51) | 82.87 (23.11) | 71.06 (32.01) | 76.54 (28.73)
  180°/s Hamstring PT/BMI(less affected knee) | 46.74 (17.76) | 56.85 (19.74) | 53.73 (22.55) | 56.76 (21.21)
  180°/s hamstring/quadriceps (less affected knee) | 0.80 (0.19) | 0.69 (0.19) | 0.76 (0.22) | 0.74 (0.18)
  60°/s Quadriceps PT/BMI(more affected knee) | 82.46 (43.96) | 118.50 (45.52) | 100.16 (47.85) | 108.06 (48.83)
  60°/s Hamstring PT/BMI(more affected knee) | 58.87 (33.60) | 77.70 (29.27) | 67.00 (30.87) | 72.80 (31.55)
  60°/s Hamstring/Quadriceps(more affected knee) | 0.77 (0.27) | 0.65 (0.12) | 0.71 (0.22) | 0.71 (0.22)
  180°/s Quadriceps PT/BMI(more affected knee) | 52.42 (25.08) | 73.62 (23.53) | 57.18 (30.59) | 62.03 (29.38)
  180°/s Hamstring PT/BMI(more affected knee) | 42.25 (25.19) | 51.38 (23.24) | 46.19 (22.20) | 48.08 (23.38)
  180°/s Hamstring/Quadriceps(more affected knee) | 0.92 (0.58) | 0.66 (0.19) | 0.94 (0.58) | 0.85 (0.48)

2. Primary Outcome: Joint Position Sense of the More and Less Affected Knees
Description: Absolute angular errors of the 15°, 45°, and 60° and the mean absolute angular error of the more and less affected knees were measured by an isokinetic dynamometer (Biodex Multijoint Pro 3) with active-active angular reproduction method. Estimating the target angel procedure was repeated at 45°, 15°, and 60° and for both the more and less affected legs. After the joint position sense testing, three angles estimated by the patients were averaged, and the angular error was calculated for each target angle. Absolute angular error was calculated by averaging the angular errors, regardless of the numbers being negative or positive. The absolute angular error values of the three target angles were averaged to obtain the mean absolute angular errors. A definite angular error value has not been defined. Literally, healthy controls and patients are compared. Higher scores indicate worser joint position sense.
Time Frame: At baseline (10 minutes before the start of the treatment) and 8 weeks after start of the treatment
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Isokinetic Exercise Baseline | Isokinetic Exercise After Treatment | Home Exercise Baseline | Home Exercise After Treatment
Number analyzed (Participants) | 19 | 19 | 21 | 21
degree
  mean absolute angular error of less affected knee | 5.56 (2.78) | 4.39 (2.32) | 5.70 (3.19) | 5.03 (2.65)
  mean absolute angular error of lmore affected knee | 4.94 (3.06) | 4.38 (1.94) | 5.76 (5.35) | 4.99 (3.59)
  15° joint position sense of less affected knee | 6.26 (4.70) | 3.87 (4.28) | 5.93 (5.26) | 5.32 (4.07)
  15° joint position sense of more affected knee | 4.61 (3.79) | 0.74 (4.04) | 4.96 (4.05) | 5.27 (3.82)
  45° joint position sense of less affected knee | 6.41 (3.61) | 5.86 (3.95) | 6.23 (4.36) | 4.94 (3.04)
  45° joint position sense of more affected knee | 4.73 (3.81) | 4.21 (2.95) | 5.80 (5.00) | 5.46 (4.62)
  60° joint position sense of less affected knee | 3.40 (3.08) | 3.39 (3.00) | 4.55 (4.78) | 3.76 (4.73)
  60° joint position sense of more affected knee | 6.02 (4.99) | 4.17 (2.52) | 4.18 (6.67) | 3.47 (3.92)

3. Primary Outcome: Tampa Scale of Kinesiophobia
Description: Kinesiophobia which is described as fear of movement and physical activity was evaluated using the Tampa Scale of Kinesiophobia, which is a 17-item self-report survey. The range of scores are from 17 to 68 where the higher scores indicate an increasing degree of kinesiophobia. If the total score was above 37 points, the patient was considered to have a high level of kinesiophobia.
Time Frame: At baseline (10 minutes before the start of the treatment) and 8 weeks after start of the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isokinetic Exercise Baseline | Isokinetic Exercise After Treatment | Home Exercise Baseline | Home Exercise After Treatment
Number analyzed (Participants) | 19 | 19 | 21 | 21
score on a scale | 42.42 (5.48) | 40.57 (7.25) | 40.33 (6.37) | 40.33 (7.72)

4. Primary Outcome: Multiple Sclerosis Quality of Life-54 Total Score, Physical and Emotional Composite Scores, and Pain Subscale Score
Description: This is a multidimensional health-related quality of life measure that combines both generic and multiple sclerosis-specific symptoms in a single instrument. The 54 items are divided into 12 multi-item and 2 single-item scales.Health distress, overall quality of life, emotional well-being, role limitations-emotional and cognitive funtion items' final scores averaged and mental composite score was calculated. Physical function, health perceptions, energy/fatigue, role limitations-physical, pain, sexual function, social function, health distress items' final scores were averaged and physical composite score was obtained.Total score was obtained by averaging the mental and physical composite scores.Final scores can be between 0-100 points for total, mental, physical and pain scores. Higher values indicate better quality of life for total, physical and mental scores and worser pain levels for pain score.
Time Frame: At baseline (10 minutes before the start of the treatment) and 8 weeks after start of the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isokinetic Exercise Baseline | Isokinetic Exercise After Treatment | Home Exercise Baseline | Home Exercise After Treatment
Number analyzed (Participants) | 19 | 19 | 21 | 21
score on a scale
  MSQoL-54 (total) | 52.20 (17.98) | 57.00 (18.95) | 61.38 (18.54) | 59.39 (20.93)
  MSQoL-54 (physical) | 50.79 (17.02) | 54.69 (18.31) | 58.64 (19.81) | 56.69 (22.10)
  MSQoL-54 (mental) | 53.59 (20.71) | 59.33 (21.81) | 64.11 (20.41) | 62.07 (22.78)
  MSQoL-54 (pain) | 54.52 (26.90) | 58.57 (30.10) | 71.74 (28.52) | 67.83 (29.94)

5. Primary Outcome: Visual Analog Scale
Description: Pain intensity was evaluated with the Visual Analog Scale. Using a ruler, a 10 cm line was drawn which provided a range of scores from 0-100. Than the patients marked the point that showed their pain intensity on this line. A higher score in Visual Analog Scale indicates greater pain intensity.
Time Frame: At baseline (10 minutes before the start of the treatment) and 8 weeks after start of the treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Isokinetic Exercise Baseline | Isokinetic Exercise After Treatment | Home Exercise Baseline | Home Exercise After Treatment
Number analyzed (Participants) | 19 | 19 | 21 | 21
score on a scale | 40.78 (34.16) | 36.68 (36.66) | 41.66 (31.11) | 42.14 (29.13)

ADVERSE EVENTS:
Time Frame: adverse events were not monitored/assessed.
Description: adverse events were not monitored/assessed.
Arm/Group | Isokinetic Exercise | Home Exercise
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The limitations of the study include the low number of patients, lower EDSS scores, lack of a long-term evaluation of isokinetic exercises, and absence of a healthy control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/24/NCT03779724/Prot_SAP_001.pdf